CLINICAL TRIAL: NCT03298126
Title: Is Conventional TR Band Deflation Protocol Inferior to Internationally Developed TR Band Removal Protocol in Reducing Occurrence of Radial Artery Occlusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Nasir Rahman, Assisstant Professor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 4402-MED-ERC-16
Record Dates: First submitted 2017-09-17; First posted 2017-10-02 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Radial Artery Occlusion
Keywords: Radial artery occlusion; TR band; Transradial catheterization
MeSH Terms: conditions — Arterial Occlusive Diseases

STUDY DESIGN:
Intervention Model Description: The parallel group, non-inferiority trial
Who Masked: Outcomes Assessor
Masking Description: Randomization was carried out after written informed consent through SNOSE (Sequentially Numbered Opaque Sealed Envelopes) method to ensure allocation concealment. Patients were randomized into two groups for TR band removal i.e. Group 1 received protocol A which is currently in practice at AKUH and group 2 underwent protocol B developed by Cohen and Alfonso which is supported by literature. The techniques for protocol A and protocol B. Radial artery patency was determined at 24 hours by a trained resident doctor who was blinded to the protocol administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR BAND Protocol A (Active Comparator): In this group, air removal from TR band was initiated after 2 hours of TR band application. 3 ml of air was removed periodically at an interval of 15 minutes until all the air is eliminated from the band. In case of bleeding or hematoma while deflating air, 4 ml of air was re-injected and observed for 30 minutes until next attempt was made to deflate the band. The data including the attempts made at deflating TR band, time and amount of air injected along with the response to each deflation i.e. occurrence of bleeding or hematoma was noted down in the proforma
  Interventions: Procedure: TR BAND removal protocol
- TR BAND PROTOCOL B (Active Comparator): In this group deflation was initiated after 2 hours of TR band application as described by Cohen and Alfonso. [6] 5 ml of air was deflated at first attempt. Next attempt was carried out after 15 minutes in which further 5 ml was removed. After 15 minutes, the remaining 2 ml of air was released from the band. In case of bleeding or hematoma at any attempt, 6 ml air was re-injected and interval for 15 minutes taken to attempt further air deflation. All the attempts and its response were recorded in the proforma filled out by the assessor.
  Interventions: Procedure: TR BAND removal protocol

INTERVENTIONS:
Procedure: TR BAND removal protocol — To assess radial artery patency after specific protocol used as already described in previous section.
  Other Names: Ultrasound doppler, plethysmography

SUMMARY:
Coronary artery disease (CAD) is one of the major health concerns among other non-communicable diseases globally. Cardiac catheterization is a diagnostic gold standard to determine the extent of disease in coronary arteries due to atherosclerosis. Among the two approaches for cardiac catheterization, trans-radial approach has gained more popularity than conventional trans-femoral approach over the past decade with availability of compression devices for radial artery that assures lesser risk of bleeding and hematoma and has translated into increased patient comfort and early mobility post procedure. Radial artery occlusion is a common complication of trans-radial procedures often ignored by the operator after procedure due to dual blood supply by ulnar artery. Although clinically silent usually, it necessitate the need of monitoring radial artery for patency because of risk of limited trans-radial access later.Reportedly, RAO occurs in about 10% of cardiac catheterizations. , compression devices applied after sheath removal may be a contributing factor to radial artery occlusion because of selective pressure for extended time duration (3-4 hours). Various protocols have been developed to remove TR band by different institutions across the globe and have been tested to assess post procedure complications. To the best of what we know, there exists no standard protocol to deflate TR band. Also, the current protocol in practice at our institution has not been evaluated against other protocols that are followed in other institution across the globe claiming lesser post procedure complications. Hence, our aim was to test through a randomized trial whether our hospital standard protocol is non-inferior to the existing international protocol of Cohen & Alfonso that promises lesser complication rate

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted for coronary angiography in specified period of study
* patients who sign informed consent

Exclusion Criteria:

* known radial artery occlusion
* > 3 radial angiograms in the past
* plan for AD- hoc PCI
* on warfarin therapy
* known bleeding diathesis or hypercoagulable state
* contraindication to radial artery access such as hemodialysis fistula, mastectomy or localized infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Radial artery occlusion (RAO) | from TR band removal upto 24 hours of hospital stay of the patient
  Radial artery patency was assessed in both groups by ultrasound doppler and bed side plethysmographic waveforms

SECONDARY OUTCOMES:
Hematoma | from TR band removal upto 24 hours of hospital stay of the patient
  Patients in both arms were assessed for the presence of hematoma in the cannulated arm used for the angiography before and after the TR band removal. Hematoma were graded from grad 1-5 according to the extent of arm involvement as per standard EASY hematoma classification system.
Re bleed | from the time of TR band application, during its removal and upto 24 hours of hospital stay of the patient
  patients in both arms were assessed for any sign of major or minor bleeding from the punctured site, such as oozing, frank bleeding which required extra pressure to apply on the site to control it, or required extra amount of air to be inflated to control it. any such event was documented as Re bleed after the TR band application.

CONTACTS AND LOCATIONS:
Overall Officials: Nasir M Rahman, FCPS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rahman N, Artani A, Baloch F, Artani M, Fatima H, Salam A, Ahmed S. Role of trans-radial band protocols in radial artery occlusion: Randomized trial. Asian Cardiovasc Thorac Ann. 2022 May;30(4):409 - 415. doi: 10.1177/02184923211027790. Epub 2021 Jun 29. PMID 34182800